CLINICAL TRIAL: NCT00005975
Title: A Phase III Trial of Placebo Versus Megestrol Acetate 20 MG/Day Versus Megestrol Acetate 40 MG/Day as Treatment for Symptoms of Ovarian Failure in Women Treated for Breast Cancer: SWOG Study S9626
Brief Title: S9626: Megestrol in Treating Hot Flashes Following Treatment for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000067962; S9626 (Other: SWOG); NCI-P00-0159 (Other: NCI); U10CA037429 (NIH)
Record Dates: First submitted 2000-07-05; First posted 2004-06-28 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; Hot Flashes
Keywords: stage I breast cancer; stage II breast cancer; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Megestrol Acetate/Placebo 20 mg/day (Active Comparator): Double blinded Megestrol Acetate 20 mg/day or Megestrol Acetate Placebo 20 mg/day taken for 3 months
  Interventions: Drug: Megestrol Acetate 20mg/day; Drug: Megestrol Acetate Placebo 20 mg/day
- Megestrol Acetate/Placebo 40 mg/day (Active Comparator): Double blinded Megestrol Acetate 40 mg/day or Megestrol Acetate Placebo 40 mg/day taken for 3 months
  Interventions: Drug: Megestrol Acetate 40 mg/day; Drug: Megestrol Acetate Placebo 40 mg/day

INTERVENTIONS:
Drug: Megestrol Acetate 20mg/day — Double blinded Megestrol Acetate 20 mg/day
  Other Names: NSC-71423
  Arms: Megestrol Acetate/Placebo 20 mg/day
Drug: Megestrol Acetate 40 mg/day — Double blinded Megestrol Acetate 40 mg/day
  Other Names: NSC-71423
  Arms: Megestrol Acetate/Placebo 40 mg/day
Drug: Megestrol Acetate Placebo 20 mg/day — Megestrol Acetate Placebo 20 mg/day
  Other Names: NSC-71423
  Arms: Megestrol Acetate/Placebo 20 mg/day
Drug: Megestrol Acetate Placebo 40 mg/day — Megestrol Acetate Placebo 40 mg/day
  Other Names: NSC-71423
  Arms: Megestrol Acetate/Placebo 40 mg/day

SUMMARY:
RATIONALE: Megestrol may be effective in treating hot flashes following treatment for breast cancer. It is not yet known which regimen of megestrol is most effective for hot flashes.

PURPOSE: Randomized phase III trial to compare the effectiveness of different doses of megestrol in treating hot flashes in patients who have undergone therapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effectiveness and duration of the benefit of placebo versus low dose megestrol versus high dose megestrol in the reduction of severe and/or frequent hot flashes in patients with previously treated invasive breast cancer. II. Document the effects of various dose levels of megestrol on atrophic vaginitis and dyspareunia in these patients. III. Evaluate the toxicity of this treatment in these patients.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to tamoxifen use (yes vs no), number of hot flashes per week (5-34 vs 35-63 vs more than 63), and duration of hot flashes (6 months or less vs longer than 6 months). Patients are randomized to one of three treatment arms. Arm I: Patients receive oral placebo daily. Arm II: Patients receive lower dose oral megestrol daily. Arm III: Patients receive higher dose oral megestrol daily. Patients who do not respond after 3 months of treatment receive an additional dose of oral megestrol daily. Treatment continues for a total of 6 months in the absence of disease progression or unacceptable toxicity. Patients are followed at 3 months.

PROJECTED ACCRUAL: A total of 279 eligible patients (93 per arm) are expected to be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of infiltrating breast cancer (T1-3, N0-1, M0) treated with appropriate local and regional therapy Chemotherapy and/or surgery completed At least 10 hot flashes per week OR At least 5 severe or very severe hot flashes per week No prior participation in NCI sponsored breast cancer adjuvant protocol No recurrent or persistent vaginal bleeding If postmenopausal and had any vaginal bleeding within past year, then must have normal endometrial biopsy Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Not specified Menopausal status: Pre or postmenopausal Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No history of deep vein thrombosis Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other prior malignancy in past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other adequately treated stage I or II cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No concurrent chemotherapy Endocrine therapy: Prior hormonal therapy allowed At least 6 months since prior megestrol At least 1 week since prior nonestrogen containing steroid hormones (except tamoxifen) Concurrent tamoxifen allowed only if begun at least 4 months prior to study No other concurrent nonestrogen containing steroid hormones No concurrent estrogen or hormone replacement therapy Radiotherapy: Concurrent radiotherapy allowed Surgery: See Disease Characteristics Prior hysterectomy allowed No concurrent surgery Other: Concurrent nonhormonal prescription or nonprescription medications for hot flashes allowed (e.g., clonidine, ergotamine tartrate, vitamin E, or soy)

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 1998-04; Primary Completion 2001-09 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness and duration of the benefit of placebo and 2 dose levels of megestrol acetate in reduction of severe and/or frequent hot flashes in patients with history of adequate local and regional treatment of invasive breast cancer | 3, 6, and 9 months

SECONDARY OUTCOMES:
Document any effects of various dose levels of megestrol acetate on atrophic vaginitis and dyspareunia | 3, 6, and 9 months
Evaluate toxicity of two dose levels of megestrol acetate relative to placebo | 3, 6, and 9 months
Feasibility of accrual patients to placebo-controlled study | At registration

CONTACTS AND LOCATIONS:
Overall Officials: John W. Goodwin, MD, Study Chair — Cancer Research for the Ozarks

REFERENCES:
- [Result] Goodwin JW, Green SJ, Moinpour CM, Bearden JD 3rd, Giguere JK, Jiang CS, Lippman SM, Martino S, Albain KS. Phase III randomized placebo-controlled trial of two doses of megestrol acetate as treatment for menopausal symptoms in women with breast cancer: Southwest Oncology Group Study 9626. J Clin Oncol. 2008 Apr 1;26(10):1650-6. doi: 10.1200/JCO.2006.10.6179. PMID 18375894